CLINICAL TRIAL: NCT02949908
Title: A Phase IV, Prospective, Multicenter, Open Label, Uncontrolled, Non-interventional, Single Arm Study to Measure Treatment Satisfaction of Multiple Sclerosis (MS) Patients on Rebif® After Discontinuing Initial First-line Treatment
Brief Title: MEasuring Satisfaction of Treatment With REbif After Initial Treatment of Multiple Sclerosis (MS)
Acronym: MESTRE-MS
Status: Terminated | Type: Observational
Why Stopped: Delay in site selection and recruitment.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck B.V., Netherlands (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200136_597
Record Dates: First submitted 2016-10-17; First posted 2016-10-31 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis; Rebif; Treatment Satisfaction Questionnaire for Medication Version II; Multiple Sclerosis International Quality of Life Questionnaire
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
  Interventions: Drug: Rebif

INTERVENTIONS:
Drug: Rebif — Participants diagnosed with RRMS who had discontinued their oral or injectable first-line multiple sclerosis (MS) medication, and have been receiving subcutaneous Interferon beta-1a (IFNβ-1b) (Rebif) were observed during the study. Participants received Rebif in accordance with the licensed Summary of Product Characteristics label or currently approved specific country product information.
  Other Names: IFNβ-1b

SUMMARY:
This is a prospective, multicenter, open label, uncontrolled, non-interventional, single arm study to measure treatment satisfaction of relapsing remitting MS (RRMS) participants on Rebif after discontinuing initial first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age (both inclusive), at the time of informed consent
* Participants diagnosed with RRMS according to McDonald criteria 2010
* Participants have discontinued treatment with dimethyl fumarate (Tecfidera), teriflunomide (Aubagio), glatiramer acetate (Copaxone®), intramuscular IFNβ-1a (Avonex®), pegylated interferon (Plegridy®), subcutaneous IFNβ-1b (Betaferon®) or fingolimod (Gilenya®) within 6 months prior to Visit 1

  * Currently treated with Rebif using RebiSmart 2.0, for a maximum of 6 months prior to Visit 1
  * Participants have a score on the Expanded Disability Status Scale (EDSS) between 0 to 5.0 inclusive
  * Participants willing and able to give informed consent.

Exclusion Criteria:

* Participants have known planned surgical procedures at the time of the informed consent that will prevent adherence to treatment with Rebif through RebiSmart 2.0
* Participants diagnosed with primary progressive, secondary progressive, or progressive relapsing MS
* pregnant or lactating, or planning to become pregnant subjects
* In the opinion of the Investigator has significant renal or hepatic impairment or other significant disease (e.g., cognitive or visual impairment) that would compromise adherence and completion of the study
* Reports any reason that he/she cannot complete the 1 year study
* Participants have a history of hypersensitivity to natural or recombinant interferon, or any other component of the formulation
* Participants who contraindicated for the treatment with subcutaneous IFNβ-1a therapy as per summary of product characteristics or currently approved specific country product information
* Participants have any other factor that in the opinion of the Investigator would make the subject unsuitable for participation in this study
* Participants have significant psychiatric symptoms that, in the opinion of the Investigator, would impact patient ability to comply with treatment recommendations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RRMS participants who have discontinued their initial MS treatment and for whom MS treatment will be required according to the decision of the Health Care Professional and participant.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck B.V., the biopharmaceutical division of Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants were enrolled and the study was prematurely terminated due to low participant recruitment.
Groups:
- Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS): Participants diagnosed with RRMS who had discontinued their oral or injectable first-line multiple sclerosis (MS) medication, and have been receiving subcutaneous Interferon beta-1a (IFNβ-1b) (Rebif) were observed during the study. Participants received Rebif in accordance with the licensed Summary of Product Characteristics label or currently approved specific country product information.
Period: Overall Study
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Study termination | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction Score Determined With Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II)
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across a wide variety of medication types and illness conditions. It consists 11 question items. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging from 1 to 7, where 1= Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied.
Time Frame: Month 6
Population: Analysis population included participant who received study medication and had data collected at Month 6.
Measure: Number; unit: Units on a scale
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 1
Units on a scale | 5

2. Primary Outcome: Treatment Satisfaction Determined With Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II)
Description: as for outcome 1
Time Frame: Month 12
Population: Data was not analyzed for this outcome as the study terminated prematurely due to low subject enrollment and no data was collected for Month 12 assessment.
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

3. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: ARR defined as the number of relapses per year. A relapse is defined as the appearance of a new clinical sign or symptom attributable to MS, or clinical worsening of a previous sign or symptom that had been stable for greater than or equal to (>=) 30 days and that persisted for >=24 hours without fever.
Time Frame: Month 12
Population: as for outcome 2
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Adherence to Treatment
Description: According to the World Health Organization (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term).
Time Frame: Month 6 and Month 12
Population: Analysis population: participant who received study medication and had data collected for evaluation. Overall Number of Participants Analyzed = those evaluable for this outcome. Number Analyzed (n) = those evaluable at specified time point and n = 0 signifies no subject was analyzed as study terminated prematurely before Month 12 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 1
Participants
  At Month 6 | 1
  At Month 12: number analyzed (Participants) | 0

5. Secondary Outcome: Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) Score at Month 6 and 12
Description: The MusiQoL is a disease-specific validated 31-item multi-dimensional, self-administered questionnaire. Participants were asked to assess their level of satisfaction with the treatment. Question was answered using a 6-point Likert scale, defined as 1-Never/Not at all, 2-Rarely/A little, 3-Sometimes/Somewhat, 4-Often/A lot, 5-Always/Very much and 6-Not applicable.
Time Frame: Month 6, Month 12
Population: as for outcome 4
Measure: Number; unit: units on a scale
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 1
units on a scale
  Month 6 | 4
  Month 12: number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Discontinued From Initial MS Treatment (Oral or Injectable) by Reason for Discontinuation
Description: Here numbers of participants who discontinued the initial MS treatment (Oral or Injectable) are reported with the reason of discontinuation.
Time Frame: Baseline
Population: Analysis population included participants who enrolled in this study and had discontinued their initial MS treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 1
Participants | 1

7. Secondary Outcome: Correlation Between Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) and Annualized Relapse Rate (ARR)
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across wide variety of medication types and illness conditions. It consists 11 question items. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging 1-7, where 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. ARR= number of relapses per year. Relapse= the appearance of a new clinical sign or symptom attributable to MS, or clinical worsening of a previous sign or symptom that had been stable for greater than or equal to (>=) 30 days and that persisted for >=24 hours without fever.
Time Frame: up to 12 months
Population: Correlation analysis was not performed because the study was terminated prematurely due to low participants recruitment (only 2 participants enrolled), which did not allow performance of the planned correlation statistical analysis.
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

8. Secondary Outcome: Correlation Between Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) and Adherence
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across wide variety of medication types and illness conditions. It consists 11 question items. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging 1-7, where 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. According to the World Health Organization (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term).
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

9. Secondary Outcome: Correlation Between Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) and Reason for Discontinuation
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across wide variety of medication types and illness conditions. It consists 11 question items. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging 1-7, where 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Reasons of discontinuation of initial MS treatment were reported.
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

10. Secondary Outcome: Correlation Between Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) and Annualized Relapse Rate (ARR)
Description: The MusiQoL is a disease-specific validated 31-item multi-dimensional, self-administered questionnaire. Participants were asked to assess their level of satisfaction with the treatment. Question was answered using a 6-point Likert scale, defined as 1-Never/Not at all, 2-Rarely/A little, 3-Sometimes/Somewhat, 4-Often/A lot, 5-Always/Very much and 6-Not applicable. ARR= number of relapses per year. Relapse= the appearance of a new clinical sign or symptom attributable to MS, or clinical worsening of a previous sign or symptom that had been stable for greater than or equal to (>=) 30 days and that persisted for >=24 hours without fever.
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

11. Secondary Outcome: Correlation Between Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) and Adherence
Description: The MusiQoL is a disease-specific validated 31-item multi-dimensional, self-administered questionnaire. Participants were asked to assess their level of satisfaction with the treatment. Question was answered using a 6-point Likert scale, defined as 1-Never/Not at all, 2-Rarely/A little, 3-Sometimes/Somewhat, 4-Often/A lot, 5-Always/Very much and 6-Not applicable. According to the World Health Organization (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term).
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

12. Secondary Outcome: Correlation Between Multiple Sclerosis International Quality of Life Questionnaire (MusiQoL) and Reason for Discontinuation
Description: The MusiQoL is a disease-specific validated 31-item multi-dimensional, self-administered questionnaire. Participants were asked to assess their level of satisfaction with the treatment. Question was answered using a 6-point Likert scale, defined as 1-Never/Not at all, 2-Rarely/A little, 3-Sometimes/Somewhat, 4-Often/A lot, 5-Always/Very much and 6-Not applicable. Reasons of discontinuation of initial MS treatment were reported.
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

13. Secondary Outcome: Correlation Between Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) Subscales and Adherence
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across wide variety of medication types and illness conditions. It consists 11 question items used for computing 4 subscales: effectiveness, convenience, side effects and global satisfaction. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging 1-7, where 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. According to the World Health Organization (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term).
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

14. Secondary Outcome: Correlation Between Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) Subscales and Reasons for Discontinuation
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across wide variety of medication types and illness conditions. It consists 11 question items used for computing 4 subscales: effectiveness, convenience, side effects and global satisfaction. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging 1-7, where 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied. Reasons of discontinuation of initial MS treatment were reported.
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

15. Secondary Outcome: Change From Baseline in Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) Subscale Score at Month 6 and Month 12
Description: TSQM v II is designed as a general measure of treatment satisfaction with medication, suitable for use across wide variety of medication types and illness conditions. It consists 11 question items used for computing 4 subscales: effectiveness, convenience, side effects and global satisfaction. Participants were asked to assess their level of satisfaction taking all things into account. Participants were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging 1-7, where 1=Extremely Dissatisfied, 2=Very Dissatisfied, 3=Dissatisfied, 4=Somewhat Satisfied, 5=Satisfied, 6=Very Satisfied, 7=Extremely Satisfied.
Time Frame: Baseline, Month 6, Month 12
Population: Data was not analyzed because study terminated prematurely due to low participant recruitment (only 2 participants enrolled). Month 6 data was available for only 1 participant and none had data collected at Month 12, which did not allow performance of planned analysis. Overall score at Month 6 was collected and is reported under primary outcome 1.
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline in Annualized Relapse Rate (ARR) at Month 12
Description: as for outcome 3
Time Frame: Baseline, Month 12
Population: as for outcome 2
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

17. Secondary Outcome: Correlation Between Annualized Relapse Rate (ARR) and Treatment Adherence
Description: ARR defined as the number of relapses per year. A relapse is defined as the appearance of a new clinical sign or symptom attributable to MS, or clinical worsening of a previous sign or symptom that had been stable for greater than or equal to (>=) 30 days and that persisted for >=24 hours without fever. According to the World Health Organization (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term).
Time Frame: up to 12 months
Population: as for outcome 7
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 7 Months
Arm/Group | Rebif in Relapsing-Remitting Multiple Sclerosis (RRMS)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to low recruitment (only 2 participants were enrolled). Therefore, no statistical analysis was performed on the limited data which was collected during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT02949908/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02949908/SAP_001.pdf